CLINICAL TRIAL: NCT00190359
Title: Modifications of the Growth Hormone/IGF1 Axis in Heart Failure Patients
Brief Title: Growth Hormone and Heart Failure
Status: Terminated | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: CRC00007
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2005-09-19 (Estimated); Status verified 2002-04

CONDITIONS: Heart Failure, Congestive
Keywords: heart failure; hormones; growth substances
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Heart failure induces modification in several neurohormonal systems. The aim of this study is to determine if the growth hormone/IGF1 axis is modified in heart failure patients compared to healthy volunteers.

DETAILED DESCRIPTION:
One hundred and sixty three heart failure patients were evaluated by clinical examination, echocardiography, exercise test and measurement of blood BNP. Growth hormone and IGF-1 plasma levels were determined in each patient. The same biological measurements were performed in a group of 148 healthy controls. Comparisons were performed between groups for Growth hormone plasma level, IGF-1 plasma level and Growth hormone/IGF-1 index. A correlation between the severity of heart failure and the different biological parameters was searched.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patients in stable condition

Exclusion Criteria:

* cancer
* pituitary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2000-09; Study Completion 2003-02

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Maison, MD, PhD, Principal Investigator — APHP